CLINICAL TRIAL: NCT00048230
Title: An International, Multi-Center, Randomized, Open-Label Study of PS-341 (VELCADE™) Versus High-Dose Dexamethasone in Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: PS-341 (VELCADE™) Versus High-Dose Dexamethasone in Patients With Relapsed or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M34101-039; NCT00052260 (obsolete NCT alias)
Record Dates: First submitted 2002-10-28; First posted 2002-10-30 (Estimated); Last update posted 2012-01-13 (Estimated); Status verified 2012-01

CONDITIONS: Multiple Myeloma
Keywords: Relapsed Multiple Myeloma; Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib

INTERVENTIONS:
Drug: bortezomib

SUMMARY:
This study will compare the efficacy of PS-341 versus high dose dexamethasone.

ELIGIBILITY:
Inclusion Criteria

* Patient is of a legally consenting age, as defined by local regulations.
* Patient is, in the investigator's opinion, willing and able to comply with the protocol requirements.
* Patient has given voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to their future medical care.
* Female patient is either post-menopausal or surgically sterilized or willing to use an acceptable method of birth control (i.e., a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study.
* Male patient agrees to use an acceptable method for contraception for the duration of the study.
* Patient was previously diagnosed with multiple myeloma based on standard criteria and currently requires second-, third-, or fourth-line therapy because of PD, defined as a 25% increase in M-protein, development of new or worsening of existing lytic bone lesions or soft tissue plasmacytomas, or hypercalcemia (serum calcium >11.5 mg/dL), or relapse from CR.
* Patient has measurable disease, defined as follows:
* For secretory multiple myeloma, measurable disease is defined as any quantifiable serum monoclonal protein value (generally, but not exclusively, greater than 1 g/dL of IgG M-Protein and greater than 0.5g/dL IgA) and, where applicable, urine light-chain excretion of ≥200 mg/24 hours.
* For oligo- or non-secretory multiple myeloma, measurable disease is defined by the presence of soft tissue (not bone) plasmacytomas as determined by clinical examination or applicable radiographs (i.e. MRI, CT-Scan). In patients with oligosecretory multiple myeloma, the serum and/or urine M-protein measurements are very low and difficult to follow for response assessments. Therefore, other disease sites (bone marrow; extramedullary mass) must be assessed and followed. In patients with non-secretory multiple myeloma, there is no M-protein in serum or urine by immunofixation.
* Patient has a Karnofsky performance status ≥60%.
* Patient has a life-expectancy >3 months.
* Patient has the following laboratory values at and within 14 days before Baseline (Day 1 of Cycle 1, before study drug administration):
* Platelet count ≥50 x 10E+9/L without transfusion support within 7 days before the laboratory test.
* Hemoglobin ≥7.5 g/dL, without transfusion support within 7 days before the laboratory test.
* Absolute neutrophil count (ANC) ≥0.75 x 10E+9/L without the use of colony stimulating factors.
* Corrected serum calcium <14 mg/dL (3.5 mmol/L).
* Aspartate transaminase (AST): ≤2.5 x the upper limit of normal (ULN).
* Alanine transaminase (ALT): ≤2.5 x the ULN.
* Total bilirubin: ≤1.5 x the ULN.
* Calculated or measured creatinine clearance: ≥20 mL/minute.

Exclusion Criteria

* Patient previously received treatment with VELCADE.
* Patient previously was refractory to treatment with high-dose dexamethasone, as experiencing less than a partial response to or PD within 6 months after discontinuing dexamethasone, or discontinued dexamethasone because of ≥Grade 3 dexamethasone-related toxicity.
* Previous high-dose dexamethasone therapy is defined as >500 mg dexamethasone or equivalent over a 10-week period, whether administered alone or as part of the VAD regimen.
* Patient received nitrosoureas within 6 weeks or any other chemotherapy, including thalidomide or clarithromycin, or radiation therapy within 3 weeks before enrollment.
* Patient received corticosteroids (>10 mg/day prednisone or equivalent) within 3 weeks before enrollment.
* Patient received immunotherapy or antibody therapy within 8 weeks before enrollment.
* Patient received plasmapheresis within 4 weeks before enrollment.
* Patient had major surgery within 4 weeks before enrollment. (Kyphoplasty is not considered major surgery.)
* Patient has a history of allergic reaction attributable to compounds containing boron or mannitol.
* Patient has peripheral neuropathy of Grade 2 or greater intensity, as defined by the NCI Common Toxicity Criteria (NCI CTC):
* Grade 2: Objective sensory loss or paresthesia (including tingling), interfering with function, but not interfering with activities of daily living (ADLs).
* Grade 3: Sensory loss or paresthesia interfering with ADLs.
* Grade 4: Permanent sensory loss that interferes with function.
* Patient had a myocardial infarction within 6 months of enrollment or has New York Heart Association (NYHA) Class III or IV heart failure uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities.
* Patient was treated for a cancer other than multiple myeloma within 5 years before enrollment, with the exception of basal cell carcinoma or cervical cancer in situ.
* Patient has cardiac amyloidosis.
* Patient has poorly controlled hypertension, diabetes mellitus, or other serious medical or psychiatric illness that could potentially interfere with the completion of treatment according to this protocol.
* Patient is known to be human immunodeficiency virus (HIV)-positive. (Patients assessed by the investigator to be at risk for HIV infection should be tested in accordance with local regulations.)
* Patient is known to be hepatitis B surface antigen-positive or has known active hepatitis C infection.
* Patient has an active systemic infection requiring treatment.
* Female patient is pregnant or breast-feeding.
* Patient currently is enrolled in another clinical research study and/or is receiving an investigational agent for any reason.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 620 (Actual)
Dates: Start 2002-06; Primary Completion 2004-07 (Actual); Study Completion 2004-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (93):
- United States (39):
  - Alta Bates Comprehensive Cancer Center, Berkeley, California
  - City of Hope, Duarte, California
  - Scripps Clinic, La Jolla, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Kaiser Permanente Oncology Clinical Trials, Vallejo, California
  - Lombardi Cancer Center, Georgetown University Medical Center, Washington D.C., District of Columbia
  - Med Star Institute, Washington Cancer Center, Washington D.C., District of Columbia
  - Hematology/Oncology Associates, PA, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - H. Lee Moffitt Cancer Center, University of S. Florida, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Northwestern University Medical School, Chicago, Illinois
  - Loyola University Medical Center: Cardinal Bernardin Cancer Center, Maywood, Illinois
  - LSU HC, Shreveport, Louisiana
  - Tufts New England Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Kirstein Room 135, Boston, Massachusetts
  - Department of Internal Medicine, Univ. of Michigan Comp. Cancer Center, Ann Arbor, Michigan
  - VA Medical Center, Sections of Hematology/Oncology, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Hackensack University Medical Center, David Jurist Research Building, Hackensack, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Long Island Jewish Medical Center, Division of Hematology/Oncology, New Hyde Park, New York
  - St. Vincent's Comprehensive Cancer Center, Research Department, New York, New York
  - NY Presbyterian Hospital, New York, New York
  - Rochester General Hospital, Lipson Cancer Blood Center, Rochester, New York
  - University of Rochester Medical Center, James P. Wilmot Cancer Center, Rochester, New York
  - Carolinas Hematology-Oncology Associates, Charlotte, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Western Pennsylvania Hospital, Dept. of Human Oncology, Pittsburgh, Pennsylvania
  - Trident Palmetto Hematology/Oncology, Charleston, South Carolina
  - Division of Hematology/Stem Cell Transplant, Nashville, Tennessee
  - Texas Oncology at Medical City Dallas Hospital, Dallas, Texas
  - Baylor Institute for Immunology Research, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Wilhelminenspital Wien, Abt. Fur Med. und Medizinische Onkologie, Vienna, Austria
- Belgium (7):
  - ACZA, Campus Stuivenberg, Antwerp
  - Institut Jules Bordet, Unite Sterile, Brussels
  - CHU Erasme / ULB University, Hematology 7th Floor, Brussels
  - C.H. Notre Dame-Reine Fabiola, Charleroi
  - UZ Gasthuisberg, Department of Hematology, Leuven
  - AZ St. Jan, Dept. of Haematology, Rugge
  - Cliniques Universitaires U.C.L de Mont Godinne, Hopital de Jour, Yvoir
- Canada (4):
  - Cross Cancer Institute, Edmonton, Alberta
  - London Health Sciences Center, London, Ontario
  - Toronto General Research Institute, Princess Margaret Hospital, Toronto, Ontario
  - Royal Victoria Hospital, Montreal, Quebec
- France (10):
  - Hospital Claude Huriez, Service des Maladies du Sang, Lille, Cedex
  - Nantes Hotel Dieu Hospital, Nantes, Cedex
  - Hopital Purpan, Pavillon Dieulafoy, Service d'Hematologie Clinique, Toulouse, Cedex
  - Institut Gustave-Roussy, Service d'Hematologie, Villejuif, Cedex
  - Hopital Antoine Beclere, Hopital de Jour de Medecine Interne, Clamart
  - Hopital Hotel Dieu, Service d'hematologie et oncologie medicale, Paris
  - Hopital Saint-Louis, Direction Financiere, Paris
  - Hopital Cochin, Service de Hematologie, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Hopital de Brabois, Service Hematologie et Medecine Interne, Vandœuvre-lès-Nancy
- Germany (12):
  - Universitatsklinikum Charite, Abt. Fuer Haematologie/Onkologie, Berlin
  - Medizinische Klinik und Poliklinik 1, Bonn
  - Universitatsklinikum Carl Gustav Carus, Dresden
  - University of Erlangen-Nurenberg, Division of Hematology/Oncology, Erlangen
  - Freiburg University Medical Center, Dept. of Hemayology/Oncology, Freiburg im Breisgau
  - Medical University Clinic (Oncology/Haematology), Hamburg
  - St. Marien Hospital, Klinik fur Hamatologie und Onkologie, Hamm
  - Universitatsklinikum Heidelberg, Abt. Fur Haematologie und Onkologie, Heidelberg
  - University of Essen Medical School, Dept. of Internal Medicine, Hufelandstr
  - Johannes Gutenberg-Universitat Mainz, III. Med Klinik und Poliknik, Mainz
  - Uniklinikum Muenster, Münster
  - Eberhard-Karls Universitat, Medizinische Klinik, Tübingen
- Belfast City Hospital, Belfast, Ireland
- Israel (2):
  - RAMBAM Medical Center, Department of Hematology and Bone, Haifa
  - Hadassah University Hospital, Jerusalem
- Italy (4):
  - Dipartmento Clinico esperimentale Di Oncologia et Ematolgia, Bergamo
  - Instituto di Ematologia e Oncologia Medica, Lorenzo e Ariosto Seragnoli, Bologna
  - Dipartimento di Biotecnologie Cellulari ed Ematologia, Roma
  - Azienda Ospedaliera, S. Giovanni Battista, Torino
- Netherlands (3):
  - Dept. of Clinical Hematology, Academic Medical Center, Amsterdam
  - Department of Hematology, Erasmus MC, 1a, Daniel Den Hoed, Rotterdam
  - Dept. Hematology, University Medical Centre, Utrecht
- Spain (2):
  - Hospital Clinico Universitario de Barcelona, Haematology Department, Barcelona
  - University Hospital of Salamanca, Salamanca
- Sweden (2):
  - Department of Haematology, Huddinge University Hospital M54, Stockholm
  - Karolinska Hospital, Dept. of Hematology, Stockholm
- United Kingdom (6):
  - Adult Leukaemia Unit, Christie Hospital, Withington, Manchester
  - Department of Haematology, Queen Elizabeth Hospital, Birmingham
  - Leeds General Infirmary, Leeds
  - Department of Haematology, St. Bartholomew's Hospital, London
  - Department of Haematology, ICSM, Hammersmith Hospital, London
  - Royal Marsden Hospital, Leukaemia and Myeloma Units, Sutton

REFERENCES:
- [Derived] Dimopoulos MA, Orlowski RZ, Facon T, Sonneveld P, Anderson KC, Beksac M, Benboubker L, Roddie H, Potamianou A, Couturier C, Feng H, Ataman O, van de Velde H, Richardson PG. Retrospective matched-pairs analysis of bortezomib plus dexamethasone versus bortezomib monotherapy in relapsed multiple myeloma. Haematologica. 2015 Jan;100(1):100-6. doi: 10.3324/haematol.2014.112037. Epub 2014 Sep 26. PMID 25261096
- [Derived] Lichter DI, Danaee H, Pickard MD, Tayber O, Sintchak M, Shi H, Richardson PG, Cavenagh J, Blade J, Facon T, Niesvizky R, Alsina M, Dalton W, Sonneveld P, Lonial S, van de Velde H, Ricci D, Esseltine DL, Trepicchio WL, Mulligan G, Anderson KC. Sequence analysis of beta-subunit genes of the 20S proteasome in patients with relapsed multiple myeloma treated with bortezomib or dexamethasone. Blood. 2012 Nov 29;120(23):4513-6. doi: 10.1182/blood-2012-05-426924. Epub 2012 Sep 27. PMID 23018640
- [Derived] van Duin M, Broyl A, de Knegt Y, Goldschmidt H, Richardson PG, Hop WC, van der Holt B, Joseph-Pietras D, Mulligan G, Neuwirth R, Sahota SS, Sonneveld P. Cancer testis antigens in newly diagnosed and relapse multiple myeloma: prognostic markers and potential targets for immunotherapy. Haematologica. 2011 Nov;96(11):1662-9. doi: 10.3324/haematol.2010.037978. Epub 2011 Jul 26. PMID 21791470
- [Derived] Vogl DT, Stadtmauer EA, Richardson PG, Sonneveld P, Schuster MW, Irwin D, Facon T, Harousseau JL, Boral A, Neuwirth R, Anderson KC. Impact of prior therapies on the relative efficacy of bortezomib compared with dexamethasone in patients with relapsed/refractory multiple myeloma. Br J Haematol. 2009 Nov;147(4):531-4. doi: 10.1111/j.1365-2141.2009.07875.x. Epub 2009 Sep 1. PMID 19725827